CLINICAL TRIAL: NCT01721408
Title: A Multicenter, Double-blind, Randomized, Comparison Study Of The Efficacy And Safety Of Tigecycline To Imipenem/Cilastatin To Treat Complicated Intra-abdominal Infections In Hospitalized Subjects.
Brief Title: A Study To Determine The Efficacy And Safety Of Tigecycline Compared With Imipenem/Cliastatin to Treat Complicated Intra-Abdominal Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1811185
Record Dates: First submitted 2012-10-31; First posted 2012-11-05 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2017-09

CONDITIONS: Intra-abdominal Infection
MeSH Terms: conditions — Intraabdominal Infections | interventions — Tigecycline; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: Tigecycline
- Group B (Active Comparator)
  Interventions: Drug: Imipenem/cilastatin

INTERVENTIONS:
Drug: Tigecycline — every 12 hours (an initial intravenous dose of 100 mg followed by 50 mg twice a day approximately every 12 hours) and placebo intravenous doses every 12 hours beginning 6 hours after the initial intravenous dose of tigecycline for at least for 5 days and up to 14 days.
  Arms: Group A
Drug: Imipenem/cilastatin — every 6 hours intravenously, and the imipenem/cilastatin will be dosed by 500mg/500mg for the subjects with creatinine clearance equal or above 71ml/min/1.73m2 or dose will be adjusted by Schedule of Study Drug Administration for Subjects with Renal Impairment.
  Arms: Group B

SUMMARY:
This is a comparative study of the efficacy and safety of tigecycline to imipenem/cilastatin in hospitalized patients with a complicated intra-abdominal infection.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized male or female subjects, at least 18 year of age.
* Complicated intra-abdominal infection is present at most under two weeks duration.
* Minimal clinical criteria at the time of intra-abdominal infection diagnosis or highly suspected intra-abdominal infection.

Exclusion Criteria:

* Anticipated length of antibiotic therapy less than 5 days or the likelihood that the subject will not complete the course of treatment.
* Intra-abdominal infection known to be caused by 1 or more bacterial pathogens not susceptible to both of the study drugs.
* Had accepted non-study antibiotics more than 24 hr within 72 hrs before enrollment except for subjects declared prior failures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (47):
- China (47):
  - Anqing City Hospital, Anqing, Anhui
  - Department of Hepatobiliary Surgery, Peking University People's Hospital, Xicheng District, Beijing Municipality
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - Department of General Surgery, the First Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of JiNan University/General Surgery, Guangzhou, Guangdong
  - The First Hospital of Shantou University School of Medicine, Shantou, Guangdong
  - Shenzhen Second People's Hosptial/Department of hepatobiliary surgery, Shenzhen, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - HaiKou Municipal People's Hospital, Haikou, Hainan
  - Hainan Provincial People's Hospital, Haikou, Hainan
  - The Third People's Hospital of Hainan Province/department of general surgery, Sanya, Hainan
  - Tongji Medical College, Huazhong University of Science and Technology, The Central Hospital of Wuhan, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University/Intensive Care Unit, Wuhan, Hubei
  - Xiangya Hospital Central-South University/General Surgery, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University/Department of General Surgery, Changsha, Hunan
  - The Third Hospital of Changsha/Department of Surgery, Changsha, Hunan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - The Affiliated Jiangyin Hospital of Southeast University Medical College, General Surgery Department, Jiangyin, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Yangzhou No.1 People's Hospital, Yangzhou, Jiangsu
  - Jilin Province People's Hospital, Changchun, Jilin
  - The First Hospital of Jilin University/Surgery, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Qinghai Provincial People's Hospital, Xining, Qinghai
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Shanghai Fengxian District Central Hospital, Department of Surgery, Shanghai, Shanghai Municipality
  - Department of General Surgery, Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - General Hospital of Chengdu Military Region of PLA, Chengdu, Sichuan
  - First people's Hospital of Kunming, Kunming, Yunnan
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang
  - Lishui People's Hospital/Intensive Care Unit, Lishui, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - China Meitan General Hospital/General Surgery Department, Beijing
  - Department of General Surgery,Beijing Shijitan Hospital,Capital Medical University, Beijing
  - Navy General Hospital PLA China/Genaral Surgery Department, Beijing
  - Peking University Third Hospital, Beijing
  - Department of General Surgery, Peking Union Medical College Hospital, Beijing
  - Institute of Antibiotics, Hua Shan Hospital, Fudan University, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Zhongshan Hospital Affiliated to Fudan University Qingpu Branch, Department of Surgery,, Shanghai
  - Tianjin Union Medical Center, Tianjin
  - Department of General Surgery, Tianjin Medical University General Hospital, Tianjin
  - Tianjin Nankai Hospital, Tianjin

REFERENCES:
- [Derived] Chen Y, Zhu D, Zhang Y, Zhao Y, Chen G, Li P, Xu L, Yan P, Hickman MA, Xu X, Tawadrous M, Wible M. A multicenter, double-blind, randomized, comparison study of the efficacy and safety of tigecycline to imipenem/cilastatin to treat complicated intra-abdominal infections in hospitalized subjects in China. Ther Clin Risk Manag. 2018 Nov 30;14:2327-2339. doi: 10.2147/TCRM.S171821. eCollection 2018. PMID 30584308
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1811185&StudyName=A%20Study%20To%20Determine%20The%20Efficacy%20And%20Safety%20Of%20Tigecycline%20Compared%20With%20Imipenem/Cliastatin%20to%20Treat%20Complicated%20Intra-Abdominal%20Infection

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the total of 470 participants randomized, 235 were randomized to each treatment group. Seven participants (4 in tigecycline group and 3 in imipenem/cilastatin group) did not receive study treatment. One participant was randomized to imipenem/cilastatin group but received tigecycline and was reported and analyzed under the tigecycline group.
Groups:
- Tigecycline 50mg: Participants were administered with tigecycline every 12 hours (an initial intravenous [IV] dose of 100 mg followed by 50 mg twice a day [BID] approximately every 12 hours) and placebo (100-mL of normal saline) IV doses every 12 hours beginning 6 hours after the initial IV dose of tigecycline.
- Imipenem/Cilastatin: Participants were administered with imipenem/cilastatin (approximately 100-mL IV infusion) intravenously approximately every 6 hours. IV placebo (100 mL of normal saline) was required to be dosed immediately After the first dose of imipenem/cilastatin.
Period: Overall Study
Arm/Group | Tigecycline 50mg | Imipenem/Cilastatin
Started | 232 (Number of participants treated.) | 231 (Number of participants treated.)
Completed | 196 | 207
Not Completed | 36 | 24
Not completed — Adverse Event | 6 | 1
Not completed — Death | 1 | 0
Not completed — Insufficient clinical response | 15 | 6
Not completed — No longer willing to participate study | 9 | 10
Not completed — Protocol Violation | 0 | 2
Not completed — Other | 3 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Does not meet entrance criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tigecycline 50mg | Imipenem/Cilastatin | Total
Number analyzed (Participants) | 232 | 231 | 463
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (18.1) | 48.2 (17.6) | 48.3 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 81 | 164
  Male | 149 | 150 | 299

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response at the Test-of-Cure (TOC) Assessment Within the Clinically Evaluable (CE) Population
Description: The clinical response was to be determined by the investigator and was classified as 1 of the following: cure (relevant clinical signs and symptoms of infection at baseline disappeared or recovered to normal and relevant non microbiological results of laboratory tests returned to normal level or the resolution of signs and symptoms so that at no further therapy was required), failure (participant required additional surgical or radiologic intervention and/or received additional anti-infection therapy to cure the infection since administration of study drug until TOC; or death after study Day 2 due to the infection or a treatment related AE or discontinuation due to a treatment related AE or received greater than 120% of the prescribed number of investigational product doses), or indeterminate (lost to follow-up; or died within 2 days after the first dose of study drug for any reason; or died after study Day 2 but prior to the TOC assessment because of non infection related reasons).
Time Frame: Day 3, Day 14 or last day of therapy (treatment duration was at least 5 days and up to 14 days), and TOC (14-21 days after the last dose of therapy)
Population: The CE population was defined as all clinical modified intent-to-treat (c-mITT) participants who satisfied clinical evaluability criteria and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tigecycline 50mg | Imipenem/Cilastatin
Number analyzed (Participants) | 207 | 205
percentage of participants
  Cure | 89.9 [84.9 to 93.6] | 96.6 [93.1 to 98.6]
  Failure | 10.1 [6.4 to 15.1] | 3.4 [1.4 to 6.9]
Statistical Analysis 1: Comparison: Tigecycline 50mg vs Imipenem/Cilastatin; Test type: Non-Inferiority or Equivalence — Assuming that the 2 treatments were equally effective, with cure rates of 75 % at the TOC assessment, the study was powered to ensure with 90% probability that the lower limit of a 2-sided 95% confidence interval (CI) for the true difference (tigecycline minus imipenem/cilastatin) in cure rates was greater than -15%; p = 0.0008, See method of CI; Difference in percentage = -6.7, 95% CI 2-sided [-12.0 to -1.4] — Used the asymptotic method corrected for continuity with normal distribution approximation. Non-inferiority test was conducted on the CE population. If non-inferiority was concluded, superiority test was conducted on both the CE and mITT populations

2. Secondary Outcome: Clinical Response at the TOC Assessment Within the Microbiologically Evaluable (ME) Population
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The ME population was defined as all CE participants who satisfied the pre-specified ME evaluable criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tigecycline 50mg | Imipenem/Cilastatin
Number analyzed (Participants) | 125 | 107
percentage of participants
  Cure | 88.0 [81.0 to 93.1] | 95.3 [89.4 to 98.5]
  Failure | 12.0 [6.9 to 19.0] | 4.7 [1.5 to 10.6]
Statistical Analysis 1: Comparison: Tigecycline 50mg vs Imipenem/Cilastatin; Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded if the lower limit of the 2-sided CI for the difference in cure rates between treatment groups (tigecycline minus imipenem/cilastatin) was greater than -15%; p = 0.0277, See method of CI; Difference in percentage = -7.3, 95% CI 2-sided [-15.2 to 0.5] — CIs and p-values for between-group treatment difference in cure rate were calculated by the asymptotic method corrected for continuity with normal distribution approximation

3. Secondary Outcome: Microbiological Response at the Subject Level in the ME Population at the TOC Assessment
Description: The microbiological response at the subject level was described according to the following definitions of efficacy. Eradication (documented or presumed): none of the baseline pathogens were present in repeat intra-abdominal cultures from the original site of infection taken during the study or a clinical response of cure precluded the necessity of a repeat intra-abdominal culture. Persistence (documented or presumed): documented: any baseline intra-abdominal pathogen was present in the cultures obtained from the original site of the intra-abdominal abscess, peritonitis, or surgical wound infection during the study; Presumed: repeat microbiological data were not obtained for a participant with a clinical response of failure. Superinfection: Emergence of a new pathogen during therapy, at the site of infection with emergence or worsening of clinical signs and symptoms of infection.
Time Frame: as for outcome 1
Population: The ME population was defined as all CE participants who satisfied the pre-specified ME evaluable criteria. n=number of participants with each microbiological response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tigecycline 50mg | Imipenem/Cilastatin
Number analyzed (Participants) | 125 | 107
percentage of participants
  Eradication (N=125, 107) | 88.0 [81.0 to 93.1] | 95.3 [89.4 to 98.5]
  Documented Eradication (N=110, 102) | 2.7 [0.6 to 7.8] | 0.0 [0.0 to 3.6]
  Presumed Eradication (N=110, 102) | 97.3 [92.2 to 99.4] | 100.0 [96.4 to 100.0]
  Persistence (N=125, 107) | 10.4 [5.7 to 17.1] | 4.7 [1.5 to 10.6]
  Documented Persistence (N=13, 5) | 7.7 [0.2 to 36.0] | 20.0 [0.5 to 71.6]
  Presumed Persistence (N=13, 5) | 92.3 [64.0 to 99.8] | 80.0 [28.4 to 99.5]
  Superinfection (N=125, 107) | 1.6 [0.2 to 5.7] | 0.0 [0.0 to 3.4]
Statistical Analysis 1: Comparison: Tigecycline 50mg vs Imipenem/Cilastatin; Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded if the lower limit of the 2-sided CI for the difference in eradication rates between treatment groups (tigecycline minus imipenem/cilastatin) was greater than -15%; p = 0.0277, See method of CI; Difference in percentage = -7.3, 95% CI 2-sided [-15.2 to 0.5] — CIs and p-values for between-group treatment difference in eradication rates were calculated by the asymptotic method corrected for continuity with normal distribution approximation

4. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) by Relationship and Seriousness
Description: An AE was any untoward medical occurrence without regard to causality in a participant who received study drug. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both AEs and Non-SAEs.
Time Frame: From the first dose of study treatment through post therapy follow-up (28 days after the last dose of therapy)
Population: Safety population included all participants who received at least 1 dose of investigational product. There was 1 participant (who was included in the safety population) had 7 AEs including 1 SAE which were identified after database release and were not reflected in the table.
Measure: Number; unit: participants
Arm/Group | Tigecycline 50mg | Imipenem/Cilastatin
Number analyzed (Participants) | 232 | 231
participants
  Number (#) of Participants with AEs | 131 | 108
  # of Participants with Treatment-Related AEs | 53 | 29
  # of Participants with SAEs | 32 | 15
  # of Participants with Treatment-Related SAEs | 19 | 7

5. Primary Outcome: Clinical Response at the TOC Assessment Within the Modified Intent-to-Treat (mITT) Population
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The MITT population was defined as all randomized participants who received at least 1 dose of investigational product.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tigecycline 50mg | Imipenem/Cilastatin
Number analyzed (Participants) | 232 | 231
percentage of participants
  Cure | 82.8 [77.3 to 87.4] | 88.7 [83.9 to 92.5]
  Failure | 10.3 [6.7 to 15.0] | 3.5 [1.5 to 6.7]
  Indeterminate | 6.9 [4.0 to 11.0] | 7.8 [4.7 to 12.0]
Statistical Analysis 1: Comparison: Tigecycline 50mg vs Imipenem/Cilastatin; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.0040, See method of CI; Difference in percentage = -6.0, 95% CI 2-sided [-12.8 to 0.8] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment (for non-serious AEs)/the time that the subject provided informed consent (for SAEs) through post therapy follow-up (28 days after the last dose of therapy)
Arm/Group | Tigecycline 50mg | Imipenem/Cilastatin
Serious Adverse Events (participants affected / at risk) | 32/232 | 16/232
Other Adverse Events (participants affected / at risk) | 57/232 | 34/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tigecycline 50mg (N=232) | Imipenem/Cilastatin (N=232)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Drug ineffective (General disorders) | 21 | 9
Sudden death (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 3 | 0
Postoperative wound infection (Infections and infestations) | 7 | 2
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Amylase increased (Investigations) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tigecycline 50mg (N=232) | Imipenem/Cilastatin (N=232)
Nausea (Gastrointestinal disorders) | 24 | 10
Vomiting (Gastrointestinal disorders) | 19 | 10
Pyrexia (General disorders) | 18 | 20
Postoperative wound infection (Infections and infestations) | 14 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.